CLINICAL TRIAL: NCT03154749
Title: Neoadjuvant Docetaxel + Carboplatin Versus Epirubicin+Cyclophosphamide Followed by Docetaxel in Triple-Negative, Early-Stage Breast Cancer (NeoCART): Study Protocol for a Multicenter, Randomized Controlled, Open-Label, Phase 2 Trial
Brief Title: DCb (Docetaxel/Carboplatin) Versus EC-D (Epirubicin/Cyclophosphamide Followed by Docetaxe) as Neoadjuvant Chemotherapy for Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Shantou Central Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Henan Cancer Hospital (Other Government); Dongguan People's Hospital (Other Government); Baotou Cancer Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170512
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Triple-Negative Breast Cancer
Keywords: Neoadjuvant chemotherapy; Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCb (Experimental): Docetaxel (75 mg/m2 administered intravenously every 3 weeks) and carboplatin (area under the concentration-time curve [AUC] 6, intravenously every 3 weeks) for six cycles
  Interventions: Drug: DCb (docetaxel/carboplatin) versus EC followed by D (epirubicin/cyclophosphamide followed by docetaxe)
- EC-D (Active Comparator): Epirubicin (90 mg/m2) plus cyclophosphamide (600 mg/m2), both administered intravenously every 3 weeks for four cycles, followed by docetaxel (100 mg/m2) administered intravenously every 3 weeks for four cycles
  Interventions: Drug: DCb (docetaxel/carboplatin) versus EC followed by D (epirubicin/cyclophosphamide followed by docetaxe)

INTERVENTIONS:
Drug: DCb (docetaxel/carboplatin) versus EC followed by D (epirubicin/cyclophosphamide followed by docetaxe) — All eligible patients were randomly assigned at a 1:1 ratio to the experimental arm (docetaxel (75 mg/m2 administered intravenously every 3 weeks) plus carboplatin (AUC 6 mg/mL per min, intravenously every 3 weeks) for six cycles) or the standard treatment arm (epirubicin (90 mg/m2) plus cyclophosphamide (600 mg/m2), both administered intravenously every 3 weeks for four cycles, followed by docetaxel (100 mg/m2) administered intravenously every 3 weeks for four cycles).

SUMMARY:
Both DCb (docetaxel/carboplatin) and EC followed by D (epirubicin/cyclophosphamide followed by docetaxe) regimens as Neoadjuvant Treatment for Triple-Negative Breast Cancer have been recommended by NCCN guideline. It is unknown which regimen is better. This study is to evaluate the efficacy and safety of DCb (docetaxel/carboplatin) and EC followed by D(epirubicin/cyclophosphamide followed by docetaxe) regimens as Neoadjuvant Treatment in Triple-Negative breast cancer. The endpoint of pathologic complete response is used as a surrogate marker for survival. Safety and tolerability assessed by number of grade 4 toxicities and hospitalizations.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) is a subtype lacking estrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor receptor type 2 (HER2) amplification. TNBC accounts for 15-20% of all invasive breast cancer. Although PARP inhibitors and immunotherapy may play a role in the treatment of early TNBC, the mainstay of treatment for TNBC is cytotoxic chemotherapy. However, despite its sensitivity to chemotherapy, TNBC is still associated with a poor prognosis.

TNBC is usually recommended for neoadjuvant therapy. The benefits of neoadjuvant therapy include reducing the size of the tumor to suit breast conserving surgery, avoiding axillary lymph node dissection, making inoperable tumors operable, and obtaining an in vivo evaluation of the tumor's chemosensitivity. Taxane- and anthracycline-based neoadjuvant regimens have become a standard treatment for TNBC, and patients have been proved to have better event-free survival (EFS) and overall survival (OS) who achieve a pathologic complete response (pCR) after neoadjuvant chemotherapy1.

Carboplatin attack cancer cells by inducing double-stranded DNA breaks, and TNBC may be sensitive to carboplatin2. Previous studies have shown that adding carboplatin to neoadjuvant chemotherapy regimens significantly improved pCR rate in TNBC patients3, 4.

Due to the long-term cardiotoxicity caused by anthracycline, several studies have explored the efficacy of neoadjuvant paclitaxel plus carboplatin regimens in TNBC and have achieved satisfactory pCR rates, but there are still controversies5. However, there is no study making comparisons between the combination of taxanes and carboplatin without anthracycline and the standard neoadjuvant regimens. Whether the combination of taxanes and carboplatin without anthracycline can achieve better efficacy while reducing adverse reactions still needs to be explored.

The NeoCART study was designed to compare the efficacy and safety of docetaxel plus carboplatin with standard neoadjuvant chemotherapy in TNBC.

ELIGIBILITY:
Eligibility Criteria：

Patients must meet the following criteria for study entry:

* Female, aged 18 Years to 70 Years
* Signed written informed consent approved by the study site Ethics Committee
* Histologically confirmed Triple-Negative invasive breast carcinoma：Pathologically confirmed as triple negative, defined as ER and PR expression both < 1 % of tumor cell nuclei per ASCO/CAP guidelinesa and HER2 negative per ASCO/CAP guidelinesa (IHC 0 or 1+ or FISH-, or IHC 2+ and FISH-)
* Stage at presentation: II - III (T1cN1-2 or T2-4N0-2)
* Patients must have measurable disease as defined by palpable lesion with caliper and/or a positive mammogram or ultrasound. Bilateral mammogram is required for study entry. Baseline measurements of the indicator lesions must be recorded on the Patient Registration Form. To be valid for baseline, the measurements must have been made within the 14 days if palpable. If not palpable, a mammogram or MRI must be done within 14 days. If palpable, a mammogram or MRI must be done within 2 months prior to study entry. If clinically indicated, x-rays and scans must be done within 28 days of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 within 14 days of study entry
* Adequate organ function within 2 weeks of study entry:

ANC ≥ 1500 cells/μL Platelet count ≥ 100,000 cells/μL Hemoglobin ≥ 9 g/dL; patients may receive red blood cell transfusions to obtain this level Serum creatinine ≤ 1.5 × upper limit of normal (ULN) INR and (activated) partial thromboplastin time (aPTT/PTT) ≤ 1.5 ×ULN AST and ALT ≤ULN Serum total bilirubin ≤ ULN, except for patients with Gilbert's syndrome for whom direct bilirubin should be within the normal range Serum alkaline phosphatase ≤ULN

* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation

Exclusion Criteria：

Patients who meet any of the following criteria will be excluded from study entry:

* Stage IV (metastatic) breast cancer
* Patients with a history of invasive breast cancer.
* Patients with a history of ductal carcinoma in situ (DCIS), except for patients treated exclusively with mastectomy > 5 years prior to diagnosis of current breast cancer
* Patients with bilateral breast cancer
* Prior chemotherapy, hormonal therapy, biologic therapy, investigational agent, targeted therapy or radiation therapy for current breast cancer.
* Patients who have undergone incisional and/or excisional biopsy of primary tumor and/or axillary lymph nodes
* History of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain disease free for greater than five years are eligible.
* Current severe, uncontrolled systemic disease that may interfere with planned treatment (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound-healing disorders)
* Major surgical procedure unrelated to breast cancer or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
* Current pregnancy and/or breastfeeding

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
PCR | Up to approximately 27-30 weeks
  Local evaluation of pCR defined as the absence of any residual invasive cancer of the resected breast specimen and all sampled ipsilateral lymph nodes (i.e., ypT0/is, ypN0 in the current AJCC staging system)

SECONDARY OUTCOMES:
Breast-conserving surgery rate | Up to approximately 27-30 weeks
  defined as the proportion of patients who achieved breast-conserving surgery out of the intent-to-treat (ITT) population of patients without inflammatory breast cancer
EFS | Up to approximately 36 months
  defined as time from randomization to disease progression, disease recurrence (local, regional, distant, or contralateral [invasive or non-invasive]), or death from any cause
OS | Up to approximately 36 months
  defined as the time from randomization to death from any cause
Adverse events | Up to approximately 27-30 weeks
  Incidence, type, and severity of all adverse events (including serious adverse events) based on NCI CTCAE, v4.0.

OTHER OUTCOMES:
Candidate predictors of pCR | Up to approximately 27-30 weeks
  BRCA, HRD, TILs，TMB, et al.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Kun, MD, Study Chair — Study Chair
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhu T, Huang YH, Li W, Wu CG, Zhang YM, Zheng XX, Zhang TF, Lin YY, Liu ZY, Ye GL, Lin Y, Wu ZY, Wang K. A non-invasive artificial intelligence model for identifying axillary pathological complete response to neoadjuvant chemotherapy in breast cancer: a secondary analysis to multicenter clinical trial. Br J Cancer. 2024 Sep;131(4):692-701. doi: 10.1038/s41416-024-02726-3. Epub 2024 Jun 25. PMID 38918556
- [Derived] Yang C, Li P, Chen Y, Zheng J, Zhang X, Gao HF, Zhang L, Wang K. Pooled analysis of NeoCARH and NeoCART trials: patient-reported outcomes in patients with early-stage breast cancer receiving platinum-based or anthracycline-based neoadjuvant chemotherapy. Support Care Cancer. 2024 Jun 3;32(6):401. doi: 10.1007/s00520-024-08610-3. PMID 38829506
- [Derived] Zhang L, Wu Z, Li J, Zhu D, Yang L, Shao Y, Lin Y, Liu Z, Cao Y, Zhang G, Shang S, Zhang Y, Wang K. Impact of Homologous Recombination Deficiency on Outcomes in Patients With Triple-Negative Breast Cancer Treated With Carboplatin-Based Neoadjuvant Chemotherapy: Secondary Analysis of the NeoCART Randomized Clinical Trial. JCO Precis Oncol. 2023 Jan;7:e2200337. doi: 10.1200/PO.22.00337. PMID 36652665
- [Derived] Li WP, Zhu T, Hu MX, Yang M, Ji F, Gao HF, Yang CQ, Zhang LL, Cheng MY, Xu FP, Wang K. Comparison of the efficacy and safety of the EC-T (epirubicin/cyclophosphamide followed by docetaxel) and TCb (docetaxel/carboplatin) neoadjuvant regimens in early TOP2A-normal stage II-III breast cancer. Neoplasma. 2020 Nov;67(6):1409-1415. doi: 10.4149/neo_2020_200130N96. Epub 2020 Jul 13. PMID 32657611